CLINICAL TRIAL: NCT02393131
Title: Neurocognitive Outcome of Conformal Whole Brain Radiotherapy With or Without Hippocampal Avoidance for Brain Metastases: A Phase II Single Blind Randomized Trial
Brief Title: Neurocognitive Outcome of Conformal WBRT w/wo Hippocampal Avoidance for Brain Metastases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201412029RINB
Record Dates: First submitted 2015-02-23; First posted 2015-03-19 (Estimated); Last update posted 2019-07-19 (Actual); Status verified 2019-03

CONDITIONS: Metastatic Malignant Neoplasm to Brain
Keywords: Brain Metastases; Whole Brain Radiotherapy; Neurocognitive function
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hippocampal avoidance WBRT (Experimental): Conformal whole brain radiotherapy with hippocampal avoidance
  Interventions: Radiation: Hippocampal avoidance WBRT
- Conformal WBRT (Active Comparator): Conformal whole brain radiotherapy without hippocampal avoidance
  Interventions: Radiation: Conformal WBRT

INTERVENTIONS:
Radiation: Hippocampal avoidance WBRT — Conformal Whole Brain Radiotherapy 30 Gy in 10 fractions with Hippocampal Avoidance using Intensity modulated radiotherapy, Volumetric arc therapy, or Tomotherapy
  Arms: Hippocampal avoidance WBRT
Radiation: Conformal WBRT — Conformal Whole Brain Radiotherapy 30 Gy in 10 fractions with Hippocampal Avoidance using Intensity modulated radiotherapy, Volumetric arc therapy, or Tomotherapy
  Arms: Conformal WBRT

SUMMARY:
Brain metastases are the most common brain tumors in adults. It is estimated that around 10-30% of cancer patients would develop brain metastases during the course of their illness.

Whole brain radiotherapy (WBRT) is the treatment of choice for the majority of patients with brain metastases. WBRT yields high radiologic response rate (27~56%) and is effective in rapid palliation of neurologic symptoms as well as prolongs time to neurocognitive function decline caused by intracranial lesions. By using conventional fractionation, 33% of patients developed late neurocognitive toxicity while memory impairment was the most common symptom. The incidence is even higher when a formal and sensitive neurocognitive assessment was prospectively evaluated. With more long-term survivors nowadays, it has become increasingly important to minimize neurocognitive function decline and maintain quality of life in patients with brain metastasis.

The function of hippocampus is cooperation in learning, consolidation and retrieval of information and essential for formation of new memories. Bilateral and unilateral radiation injury of the hippocampus is known to alter learning and memory formation. Several preclinical studies support the hypothesis of hippocampus-mediated cognitive dysfunction by ionizing radiation. Clinical studies show increase in radiation dose to hippocampus is associated with subsequent neurocognitive function impairment in adult and pediatric patients. Furthermore, the preliminary result of Radiation Therapy Oncology Group (RTOG) 0933 suggested hippocampal avoidance significant reduce the mean relative decline at 4 months from 30% in historical cohort with WBRT to 7% in experimental cohort.

Previous studies showed brain structures other than hippocampus are also associated with radiation-induced decline in neurocognitive function. There is presence of placebo effect for interventions seeking improvement in neurocognitive function. In present study, a single blind randomized phase II trial is designed to investigate the effectiveness of neurocognitive function preservation using conformal WBRT with or without hippocampal avoidance.

DETAILED DESCRIPTION:
This is a single institutional, randomized phase II study to assess the neurocognitive outcome of conformal WBRT with or without hippocampal avoidance in patients with multiple brain metastases.

Patients will be randomly assigned 1:1 to receive conformal WBRT with or without hippocampal avoidance using permuted blocks within strata that are defined by Graded Prognostic Assessment (GPA) score and baseline neurocognitive status. All patients and co-investigators except the principal investigator and attending radiation oncologists will be blinded for treatment groups.

The whole brain planning target volume (PTV) will receive 30 Gy in 10 fractions. Treatment will be delivered once daily, 5 fractions per week, over 2 to 2.5 weeks. Breaks in treatment should be minimized.

Hippocampal Avoidance WBRT:

The dose is prescribed such as 90% of cranial content PTV is covered by the prescription dose.

Maximum dose to 2% of the PTV (D2%) is 37.5 Gy, and minimum dose to 98% of the PTV (D98%) is 25 Gy. Minimum dose to 100% of the hippocampal avoidance regions is 10 Gy, and dose to any point within the hippocampal avoidance regions cannot exceed 17 Gy.

Conformal WBRT:

The dose is prescribed such as 95% of cranial content PTV is covered by the prescription dose.

Maximum dose to 1% of the PTV (D1%) is 36 Gy, and minimum dose to 99% of the PTV (D99%) is 27 Gy.

Follow-up & Assessment

Side effect evaluation:

* Acute (≤ 90 days from WBRT start) toxicities (CTCAE ver.4)
* Late (> 90 days from WBRT start) toxicities (CTCAE ver.4)

Functional evaluation: at baseline, 2-, 4- ,and 6-month, every 3 months for 12 months until intracranial disease progression or death after WBRT

* Neurocognitive function
* Self-reported cognitive functioning (two items from EORTC Quality of Life Questionnaire-C30 Taiwan)
* Health-related quality of life specific for brain neoplasms (EORTC Quality of Life Questionnaire-Brain Neoplasm Taiwan)

Efficacy evaluation:

* Follow-up brain MRI at 4-, 9- ,and 12-month until intracranial disease progression, or death.
* Overall survival

ELIGIBILITY:
Inclusion criteria:

To be eligible for inclusion, patients must fulfill the following criteria:

1. Patients with a histologic diagnosis of non-hematopoietic malignancy and radiographic evidence of brain metastases
2. Patients with brain metastasis outside a 5-mm margin around either hippocampus on gadolinium contrast enhanced MRI obtained within 30 days prior to registration
3. Patients with brain metastasis who have not been or will not be treated with stereotactic radiosurgery (SRS) or have ￼￼received SRS for￼≤ 5 intracranial ￼metastatic ￼lesions
4. No evidence of leptomeningeal metastasis on gadolinium-enhanced MRI within 30 days prior registration
5. Age ≥ 20 years
6. Karnofsky Performance Status ≥ 60%
7. Life expectancy of ≥ 4 months.
8. Women of childbearing potential and male participants must practice adequate contraception
9. Patients must be able to comply with the study protocol and follow-up schedules and provide study- specific informed consent

Exclusion criteria:

Patients fulfill any of the following criteria will be excluded from this trial

1. Prior radiotherapy to brain or SRS to > 5 intracranial metastatic lesion(s) or the biological equivalent dose in 2-Gy fractions was greater than 7.3 Gy to 40% of the volume of bilateral hippocampus from prior SRS
2. Serum creatinine > 2.0 mg/dL within 30 days prior registration
3. Contraindication to MRI such as implanted metal devices or foreign bodies, severe claustrophobia
4. Patients with leptomeningeal metastases
5. Severe, active comorbidities which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and adverse events of the protocol, or limit compliance with study requirements, defined as follows:

   1. Uncontrolled active infection requiring intravenous antibiotics at the time of registration
   2. Transmural myocardial infarction ≤ 6 months prior to registration
   3. Unstable angina or congestive heart failure requiring hospitalization ≤ 6 months prior to registration
   4. Life-threatening uncontrolled clinically significant cardiac arrhythmias
   5. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
   6. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
   7. Uncontrolled psychiatric disorder
   8. Uncontrolled, clinically significant cardiac arrhythmias
6. Will receive any other investigational agent or chemotherapy and/or target therapies during WBRT
7. Women of childbearing potential and male participants who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the radiation treatment involved in this study may be significantly teratogenic

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-03-03 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Hopkins Verbal Learning Test-Revised (HVTL-R) delayed recall score | At 4 months after radiotherapy
  Decline in Hopkins Verbal Learning Test-Revised (HVTL-R) delayed recall score from baseline to 4 months after the start of conformal whole brain radiotherapy with or without hippocampal avoidance for brain metastases

SECONDARY OUTCOMES:
Neurocognitive function by a standardized neurocognitive battery | at 1, 2, 4, 6, 9, 12 months after radiotherapy, and then every 3 months until date of death from any cause, assessed up to 24 months
  Evaluate neurocognitive function by a standardized neurocognitive battery (HVTL-R, Trail Making Test Part A & B, forward & backward Digit Span).
Patient reported outcome (Quality of Life questionnaire) | at 1, 2, 4, 6, 9, 12 months after radiotherapy, and then every 3 months until date of death from any cause, assessed up to 24 months
  EORTC Quality of Life-Core 30 questionnaire module and Quality of Life questionnaire -brain
Acute toxicity (Common Toxicity Criteria for Adverse Events version 4) | From date of radiotherapy until 90 days after radiotherapy starts
  Common Toxicity Criteria for Adverse Events version 4
Late toxicity (Common Toxicity Criteria for Adverse Events version 4) | From 90 days after radiotherapy starts until the date of death from any cause, up to 60 months
  Common Toxicity Criteria for Adverse Events version 4
Intracranial progression (Number of participant with intracranial progression on MRI of brain) | From date of enrolment until the date of first documented intracranial progression or date of death from any cause, whichever came first, assessed up to 60 months
  Number of participant with intracranial progression on MRI of brain
Overall survival | From date of enrollment until the date of death from any cause, assessed up to 60 months
  Number of patients died

OTHER OUTCOMES:
Genomic risk of neurocognitive decline after WBRT | At 4 months after radiotherapy
  Number of participants with Genomic risk of neurocognitive impairment after WBRT

CONTACTS AND LOCATIONS:
Overall Officials: Feng-Ming Hsu, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang WC, Chen YF, Yang CC, Wu PF, Chan HM, Chen JL, Chen GY, Cheng JC, Kuo SH, Hsu FM. Hippocampal avoidance whole-brain radiotherapy without memantine in preserving neurocognitive function for brain metastases: a phase II blinded randomized trial. Neuro Oncol. 2021 Mar 25;23(3):478-486. doi: 10.1093/neuonc/noaa193. PMID 32789503